CLINICAL TRIAL: NCT01024647
Title: Optimizing Response in Crohn's Disease Patients Who Have Insufficient Initial Response or Who Have Loss of Successful Response to Certolizumab Pegol (Cimzia) Induction Therapy
Brief Title: Optimizing Cimzia in Crohn's Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlanta Gastroenterology Associates (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Douglas C. Wolf, MD, Medical Director of Clinical Research, Atlanta Gastroenterology Associates
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMZ-2010
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Loss of Reponse Reinduction Responders (Active Comparator): Loss of Response Reinduction Responders:certolizumab pegol (Cimzia) 200 mg every 2 weeks
  Interventions: Biological: certolizumab pegol
- Response loss Reinduction Non-Responders (Active Comparator): Response Loss Reinduction Non-Responders:certolizumab pegol(Cimzia) 400 mg every 2 weeks
  Interventions: Biological: certolizumab pegol
- Responders (Active Comparator): Responders: certolizumab pegol(Cimzia) 400 mg every 4 weeks
  Interventions: Biological: certolizumab pegol
- Non-Responders (Active Comparator): Non-Responders: certolizumab pegol (Cimzia) 400 mg every 2 weeks
  Interventions: Biological: certolizumab pegol

INTERVENTIONS:
Biological: certolizumab pegol — certolizumab pegol 200 mg every 2 weeks
  Other Names: Cimzia
  Arms: Loss of Reponse Reinduction Responders
Biological: certolizumab pegol — certolizumab pegol 400 mg every 2 weeks
  Other Names: Cimzia
  Arms: Response loss Reinduction Non-Responders
Biological: certolizumab pegol — certolizumab pegol 400 mg every 4 weeks
  Other Names: Cimzia
  Arms: Responders
Biological: certolizumab pegol — certolizumab pegol 400 mg every 2 weeks
  Other Names: Cimzia
  Arms: Non-Responders

SUMMARY:
The purpose of this study is to determine if increasing the dose and/or dosing frequency of certolizumab pegol (Cimzia) is effective in regaining and optimizing response in patients with moderate to severe Crohn's disease.

DETAILED DESCRIPTION:
This open label study for patients with moderate to severe Crohn's disease will evaluate treatment options to improve capture of initial response and to regain loss of response to certolizumab pegol (Cimzia). It is a 26 week open label clinical trial that may be extended to 52 weeks in patients who respond to treatment during the initial 26 week study. The following dosing options will be tested: 1) Re-induction (one supplemental dose of 400mg) 2) Dose splitting (200mgQ2W) and 3) Dose Escalation (400mg Q2W. The highest dose in the study, 400mg Q2W, has been used in a large phase III trial (WELCOME) without any new safety signals. Efficacy and safety measures will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* ileal and/or colonic Crohn's disease
* moderate to severe Crohn's disease

Exclusion Criteria:

* short bowel syndrome
* ostomy
* anti-TNF therapy within 4 weeks
* prior certolizumab therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index | 26 Weeks, if responder up to 52 weeks
  ≥ 100 point decrease in CDAI represents response

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Wolf, MD, Principal Investigator — Atlanta Gastroenterology Associates
Locations (1):
- Atlanta Gastroenterology Associates, Atlanta, Georgia, United States